CLINICAL TRIAL: NCT00173888
Title: A Randomized Phase II Study of Weekly Docetaxel Plus Cisplatin Followed by Gemcitabine Versus Gemcitabine Plus Cisplatin Followed by Weekly Docetaxel in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Docetaxel Plus Cisplatin Followed by Gemcitabine Versus Gemcitabine Plus Cisplatin Followed by Docetaxel for Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 920303
Record Dates: First submitted 2005-09-08; First posted 2005-09-15 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Combination, Chemotherapy,non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Docetaxel, Cisplatin
- B (Active Comparator)
  Interventions: Drug: Gemcitabine, Cisplatin

INTERVENTIONS:
Drug: Docetaxel, Cisplatin — docetaxel 36mg/m2 IF 30 mins on day 1,8,15 cisplatin 75mg/m2 IF 2 hrs on day 15
  Arms: A
Drug: Gemcitabine, Cisplatin — gemcitabine 1000mg/m2 IF 30mins on D 1,8,15, cisplatin 75mg/m2 IF 2 hrs on day 15
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the 1-year treatment failure rate of two sequential chemotherapy regimens: weekly docetaxel plus cisplatin followed by gemcitabine; and gemcitabine plus cisplatin followed by weekly docetaxel。

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in men and women worldwide. Shifting trends in the incidence of lung cancer closely follow the patterns of cigarette smoking, although other carcinogens have been implicated. Despite intensive treatment over the past several decades, the 5-year lung-cancer survival rate remains a dismal 8-14%.

Chemotherapy is the primary therapy to patients with stage IIIB/IV disease, and most investigators believe that treatment with a combination of two agents is the best first-line treatment for stage IV NSCLC. In the late 1970s and 1980s, studies were conducted using combinations of agents. Outcomes were improved and these agents were eventually incorporated into clinical practice.

Weekly docetaxel is being studied in combination with other commonly used NSCLC chemotherapeutic agents including carboplatin, navelbine, and gemcitabine. These combinations are being studied in both first- and second-line settings. Second line chemotherapy with docetaxel may affect survival (TAX 318, 1 year survival 37% vs. 11%). However, the optimal sequence of chemotherapy was rarely explored. Weekly docetaxel may offer better tolerability vs. 3-weekly schedule when combining docetaxel to cisplatin. Based upon these studied, we choose weekly docetaxel in combination with cisplatin as our regimen. We expected the regimen would be effective and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage IIIB/IV NSCLC, no prior chemotherapy
* Age > 18 years and < 75 years
* WHO PS: 0,1
* Unidimensional or bi-dimensional measurable disease
* Neutrophils > 1.5 109/l, Platelets > 100 109/l, Hemoglobin > 10g/dl, Total bilirubin < 1.5 UNL, AST (SGOT) and ALT (SGPT) < 2.5 UNL, Alkaline phosphatases < 5 UNL; except in presence of only bone metastasis and in the absence of any liver disorders
* Creatinine < 1 UNL, and creatinine clearance should be > 60 ml/min.
* Life expectancy > 12 weeks

Exclusion Criteria:

* Pregnant, or lactating patients
* Known clinical brain or leptomeningeal involvement
* Pre-existing motor or sensory neurotoxicity of a severity > grade 1 by NCIC-CTG criteria
* CHF, angina or arrhythmias
* History of significant neurological or psychiatric disorders
* Active uncontrolled infection
* Contraindication for the use of corticosteroids
* Concurrent treatment with other experimental drugs within 30 days prior to study entry
* Concurrent treatment with any other anti-cancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the 1-year treatment failure rate of two sequential chemotherapy regimens. | 2003~2009

SECONDARY OUTCOMES:
To evaluate the response rate for each regimen, the toxicity of each arm, and the duration of response | 2003~2009

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, M.D.,Ph.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital; Ann-Lii Cheng, M.D.,Ph.D., Study Chair — Department of Oncology , National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan